CLINICAL TRIAL: NCT06166602
Title: Comparison of the Impacts of Ultrasound-guided Pericapsular Nerve Group (PENG) Block Applied in Different Volumes on Postoperative Pain in Hip Replacement Surgeries: A Randomized Clinical Trial
Brief Title: US-guided Pericapsular Nerve Group (PENG) Block in Different Volumes on Postoperative Pain in Hip Replacement Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gokce Alis, Principal Investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/0455
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Regional Anesthesia; Postoperative Pain; Hip Surgery
Keywords: Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator is not masked as different volumes are applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): PENG block was planned to be applied to group 1 patients with 20 cc of 0.25% bupivacaine.
  Interventions: Drug: PENG block with 0.25% bupivacaine.
- Group 2 (Active Comparator): PENG block was planned to be applied to group 2 patients with 10 cc of 0.25% bupivacaine.
  Interventions: Drug: PENG block with 0.25% bupivacaine.

INTERVENTIONS:
Drug: PENG block with 0.25% bupivacaine. — Peng block will be applied to the same side as the surgery, using 0.25% bupivacaine at the same concentration in different volumes.
  Other Names: Marcain®

SUMMARY:
Postoperative pain management has an important place in anesthesia practices. In order to ensure patient comfort after the surgery, to start postoperative rehabilitation early, and to prevent the process from causing mood disorders such as anxiety and pathological conditions such as chronic pain syndrome, the pain caused by the operation in the postoperative period must be effectively relieved. Pericapsular nerve group (PENG) block; It is a regional anesthesia technique that targets the anterior capsule of the hip joint and aims to block the joint branches of the accessory obturator nerve and femoral nerve by administering local anesthetic. Although it has been described recently, controlled prospective studies in the literature have shown it to be a safe and effective regional technique for postoperative pain after hip surgery. However, volume studies on this block are limited.

Therefore, in this study, we aimed to determine the optimal dose by comparing the effectiveness of PENG block on pain using different local anesthetic volumes.

DETAILED DESCRIPTION:
Postoperative pain management has an important place in anesthesia practices. In order to ensure patient comfort after the surgery, to start postoperative rehabilitation early, and to prevent the process from causing mood disorders such as anxiety and pathological conditions such as chronic pain syndrome, the pain caused by the operation in the postoperative period must be effectively relieved. Pericapsular nerve group (PENG) block; It is a regional anesthesia technique that targets the anterior capsule of the hip joint and aims to block the joint branches of the accessory obturator nerve and femoral nerve by administering local anesthetic. Although it has been described recently, controlled prospective studies in the literature have shown it to be a safe and effective regional technique for postoperative pain after hip surgery. However, volume studies on this block are limited.

Therefore, in this study, we aimed to determine the optimal dose by comparing the effectiveness of PENG block on pain using different local anesthetic volumes

It was planned to be performed with patients who had hip replacement surgery and patients who are included in the study after obtaining the necessary consents will be randomly assigned to one of Group I or Group II by sealed envelope method. Patients taken to the operating room will receive standard monitoring such as ECG, peripheral oxygen saturation and noninvasive blood pressure monitoring. Midazolam 1 mg IV, fentanyl 1 mcg/kg IV, propofol 1.5-2 mg/kg IV and rocuronium 0.6 mg/kg IV. After routine anesthesia induction, the patient will be intubated with the appropriate intubation tube. Anesthesia maintenance will be provided with 0.8 MAC sevoflurane and remifentanil infusion, as we apply in our routine. Ventilator parameters will be regulated as FiO2 50%, Vt: 0.8 ml/kg, and respiratory frequency 10-14/min, so that EtCO2 is in the range of 25-40 mmHg. Near the end of the operation, our routine analgesic application is 0.1mg/kg IV Morphine will be administered. After the operation is completed, the pericapsular nerve group block will be performed by entering the patient's suprainguinal area with a 100 mm block needle under ultrasound guidance, as in the standard practice of our clinic, and local anesthetic will be administered to the area between the psoas muscle tendon and the hip joint. During the procedure, ultrasound will be used to determine the location and visualize the distribution of the administered drug. The administered drug volume was planned to be 20 cc of 0.25% bupivacaine for group I patients and 10cc of 0.25% bupivacaine for group II patients (their concentrations would be the same but their volumes would be different). Then, the patient will be awakened from anesthesia; Patients with adequate respiratory effort below sevoflurane 0.2 MAC should receive atropine 0.1 mg/kg and neostigmine 0.05 mg/kg IV, which we routinely use, will be applied and extubated. Postoperative 30th minute, 4th hour, 6th hour, 12th hour, 24th hour pain intensities of the patients were evaluated using NRS (Numerical rating Scale) score (0-10) and postoperative Nausea and Vomiting Descriptive Scale (0 = none, 1 = mild nausea, 2 = nausea, 3 = vomiting once, 4 = vomiting more than once) will be evaluated and recorded. At the end of the surgery, patients will be given IV Morphine PCA (patient controlled analgesia) with a 2 ml bolus at a concentration of 0.5 mg/cc for 15 minutes and the amount of Morphine used during the hours when the patient's NRS score is recorded will be recorded. The patients' mobilization time after the operation will be recorded. 0.15 mg/kg IV Ondansetron will be administered for patients with Postoperative Nausea and Vomiting Descriptive Scale 2 and above. 24 hours after the surgery, patient satisfaction will be evaluated and recorded on a Likert Satisfaction scale (1-5).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with informed consent
2. Patients planned for hip surgery
3. Those between the ages of 18-80
4. ASA (American Society of Anesthesiologists) I-III patients

Exclusion Criteria:

1. Patients who do not give consent
2. Patients with coagulopathy
3. Patients with a history of local anesthetic drug allergy and toxicity
4. Patients with advanced organ failure
5. Patients with mental retardation
6. Patients with infection at the injection site
7. Pediatric patients and patients over 80 years of age
8. Pregnant patients will not be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale Score | Up to 24 hours
  Numeric Rating Scale Score (0: No pain, 10: Worst pain imaginable)

SECONDARY OUTCOMES:
Postoperative Opioid Consumption | Up to 24 hours
  24 hour morphine consumption on PCA device
Postoperative Nausea and Vomiting | Up to 24 hours
  Postoperative Nausea and Vomiting Scale (0: no PONV, 1: mild nausea, 2: severe nausea, 3: vomiting once in 24 hours, 4: Vomiting more than once in 24 hours)
Patient satisfaction | Up to 24 hours
  Likert scale (1-5, 1: very unsatisfied, 2: unsatisfied, 3: neutral, 4: satisfied, 5: very satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Choi YS, Park KK, Lee B, Nam WS, Kim DH. Pericapsular Nerve Group (PENG) Block versus Supra-Inguinal Fascia Iliaca Compartment Block for Total Hip Arthroplasty: A Randomized Clinical Trial. J Pers Med. 2022 Mar 6;12(3):408. doi: 10.3390/jpm12030408. PMID 35330408
- [Background] Lin DY, Brown B, Morrison C, Fraser NS, Chooi CSL, Cehic MG, McLeod DH, Henningsen MD, Sladojevic N, Kroon HM, Jaarsma RL. The Pericapsular Nerve Group (PENG) block combined with Local Infiltration Analgesia (LIA) compared to placebo and LIA in hip arthroplasty surgery: a multi-center double-blinded randomized-controlled trial. BMC Anesthesiol. 2022 Aug 6;22(1):252. doi: 10.1186/s12871-022-01787-2. PMID 35933328